CLINICAL TRIAL: NCT02971176
Title: Low-dose Protocol for Computed Tomography-guided Lung Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xuzhou Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 20161115-010
Record Dates: First submitted 2016-11-17; First posted 2016-11-22 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Lung Cancer, Adenocarcinoma; Lung Inflammatory Pseudotumor
MeSH Terms: conditions — Adenocarcinoma of Lung; Plasma Cell Granuloma, Pulmonary

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-dose protocol (Experimental): Patients undergo low-dose protocol computed tomography-guided lung biopsy on day 1.
  Interventions: Radiation: Low-dose protocol computed tomography
- Standard-dose protocol (Active Comparator): Patients undergo standard-dose protocol computed tomography-guided lung biopsy on day 1.
  Interventions: Radiation: Standard-dose protocol computed tomography

INTERVENTIONS:
Radiation: Low-dose protocol computed tomography — Radiation dose under the low-dose protocol computed tomography (120 kilovolt, 15 milliampere seconds)
  Arms: Low-dose protocol
Radiation: Standard-dose protocol computed tomography — Radiation dose under the standard-dose protocol computed tomography (120 kilovolt, 150 milliampere seconds)
  Arms: Standard-dose protocol

SUMMARY:
The purpose of this study is to compare the diagnostic accuracy and complication rate between low-dose computed tomography-guided and standard-dose computed tomography-guided lung biopsy.

DETAILED DESCRIPTION:
With the comprehensive usage of computed tomography examination, patients are more and more aware of the radiation dose of computed tomography. Concerns over the potential for radiation induced malignancies have increasingly been published in the scientific literature and reported in the popular press. The risk is highest for younger patients, who have more radiation-sensitive tissues and longer life expectancies than adults. Recently, the United States Food and Drug Administration announced an initiative to reduce unnecessary radiation exposure from medical imaging. At present, low-dose computed tomography protocol is widely used for the diagnosis of cardiovascular and cerebrovascular diseases.

Computed tomography-guided lung biopsy is widely used for diagnosis of lung nodules and masses. However, it requires repeating scanning to guide the needles, which inevitably increases the radiation dose. Therefore, low-dose protocol was also used in the computed tomography-guided lung biopsy procedure.

The purpose of this study is to compare the diagnostic accuracy and complication rate between low-dose computed tomography-guided and standard-dose computed tomography-guided lung biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Non-diagnostic lung lesions; Solid lung lesions; Lesion size ≥ 5mm.

Exclusion Criteria:

* The lesion which has been punctured previously; Severe dysfunction in heart, lung and coagulation function.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | From the date of randomization until the date of first documented final diagnosis, assessed up to 24 months
  Diagnostic accuracy is defined as the biopsy diagnosis matches with the final diagnosis. The final diagnosis is made according to the surgical or follow-up findings.

SECONDARY OUTCOMES:
Complication | From the date of randomization until the date of first documented biopsy-related complication, assessed up to 1 day.
  Biopsy-related complications mainly include pneumothorax and hemoptysis. Complications is evaluated by computed tomography scan and clinical symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Zi-Qi Tao, MD, Principal Investigator — Science and Education Division of Xuzhou Central Hospital
Locations (1):
- Xuzhou Central Hospital, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available.

REFERENCES:
- [Background] Fazel R, Krumholz HM, Wang Y, Ross JS, Chen J, Ting HH, Shah ND, Nasir K, Einstein AJ, Nallamothu BK. Exposure to low-dose ionizing radiation from medical imaging procedures. N Engl J Med. 2009 Aug 27;361(9):849-57. doi: 10.1056/NEJMoa0901249. PMID 19710483
- [Background] Brenner DJ, Hall EJ. Computed tomography--an increasing source of radiation exposure. N Engl J Med. 2007 Nov 29;357(22):2277-84. doi: 10.1056/NEJMra072149. No abstract available. PMID 18046031
- [Background] Jaffe TA, Yoshizumi TT, Toncheva G, Anderson-Evans C, Lowry C, Miller CM, Nelson RC, Ravin CE. Radiation dose for body CT protocols: variability of scanners at one institution. AJR Am J Roentgenol. 2009 Oct;193(4):1141-7. doi: 10.2214/AJR.09.2330. PMID 19770340
- [Background] Gnannt R, Winklehner A, Goetti R, Schmidt B, Kollias S, Alkadhi H. Low kilovoltage CT of the neck with 70 kVp: comparison with a standard protocol. AJNR Am J Neuroradiol. 2012 Jun;33(6):1014-9. doi: 10.3174/ajnr.A2910. Epub 2012 Feb 2. PMID 22300930
- [Background] Zhang LJ, Qi L, De Cecco CN, Zhou CS, Spearman JV, Schoepf UJ, Lu GM. High-pitch coronary CT angiography at 70 kVp with low contrast medium volume: comparison of 80 and 100 kVp high-pitch protocols. Medicine (Baltimore). 2014 Nov;93(22):e92. doi: 10.1097/MD.0000000000000092. PMID 25396334
- [Background] Neefjes LA, Dharampal AS, Rossi A, Nieman K, Weustink AC, Dijkshoorn ML, Ten Kate GJ, Dedic A, Papadopoulou SL, van Straten M, Cademartiri F, Krestin GP, de Feyter PJ, Mollet NR. Image quality and radiation exposure using different low-dose scan protocols in dual-source CT coronary angiography: randomized study. Radiology. 2011 Dec;261(3):779-86. doi: 10.1148/radiol.11110606. Epub 2011 Oct 3. PMID 21969666
- [Background] Chen GZ, Zhang LJ, Schoepf UJ, Wichmann JL, Milliken CM, Zhou CS, Qi L, Luo S, Lu GM. Radiation dose and image quality of 70 kVp cerebral CT angiography with optimized sinogram-affirmed iterative reconstruction: comparison with 120 kVp cerebral CT angiography. Eur Radiol. 2015 May;25(5):1453-63. doi: 10.1007/s00330-014-3533-y. Epub 2015 Jan 31. PMID 25636415
- [Background] Nour-Eldin NE, Alsubhi M, Emam A, Lehnert T, Beeres M, Jacobi V, Gruber-Rouh T, Scholtz JE, Vogl TJ, Naguib NN. Pneumothorax Complicating Coaxial and Non-coaxial CT-Guided Lung Biopsy: Comparative Analysis of Determining Risk Factors and Management of Pneumothorax in a Retrospective Review of 650 Patients. Cardiovasc Intervent Radiol. 2016 Feb;39(2):261-70. doi: 10.1007/s00270-015-1167-3. Epub 2015 Jul 7. PMID 26148648
- [Background] Nour-Eldin NE, Alsubhi M, Naguib NN, Lehnert T, Emam A, Beeres M, Bodelle B, Koitka K, Vogl TJ, Jacobi V. Risk factor analysis of pulmonary hemorrhage complicating CT-guided lung biopsy in coaxial and non-coaxial core biopsy techniques in 650 patients. Eur J Radiol. 2014 Oct;83(10):1945-52. doi: 10.1016/j.ejrad.2014.06.023. Epub 2014 Jul 5. PMID 25063212
- [Background] Kallianos KG, Elicker BM, Henry TS, Ordovas KG, Nguyen J, Naeger DM. Instituting a Low-dose CT-guided Lung Biopsy Protocol. Acad Radiol. 2016 Sep;23(9):1130-6. doi: 10.1016/j.acra.2016.05.013. Epub 2016 Jun 14. PMID 27317393
- [Background] Adiga S, Athreya S. Safety, efficacy, and feasibility of an ultra-low dose radiation protocol for CT-guided percutaneous needle biopsy of pulmonary lesions: initial experience. Clin Radiol. 2014 Jul;69(7):709-14. doi: 10.1016/j.crad.2014.02.006. Epub 2014 Apr 4. PMID 24709093
- [Background] Smith JC, Jin DH, Watkins GE, Miller TR, Karst JG, Oyoyo UE. Ultra-low-dose protocol for CT-guided lung biopsies. J Vasc Interv Radiol. 2011 Apr;22(4):431-6. doi: 10.1016/j.jvir.2011.01.431. PMID 21463754
- [Background] Meng XX, Kuai XP, Dong WH, Jia NY, Liu SY, Xiao XS. Comparison of lung lesion biopsies between low-dose CT-guided and conventional CT-guided techniques. Acta Radiol. 2013 Oct;54(8):909-15. doi: 10.1177/0284185113485937. Epub 2013 Jul 1. PMID 23817682
- [Derived] Fu YF, Li GC, Xu QS, Shi YB, Wang C, Wang T. Computed tomography-guided lung biopsy: a randomized controlled trial of low-dose versus standard-dose protocol. Eur Radiol. 2020 Mar;30(3):1584-1592. doi: 10.1007/s00330-019-06464-6. Epub 2019 Nov 27. PMID 31776740